CLINICAL TRIAL: NCT04582539
Title: A Phase 1/2, Open-Label, Multicenter Study of INCB000928 Administered as a Monotherapy in Participants With Anemia Due to Myelodysplastic Syndromes or Multiple Myeloma
Brief Title: To Assess the Safety and Tolerability of INCB000928 in Participants With Myelodysplastic Syndromes or Multiple Myeloma
Acronym: LIMBER
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic Business Decision
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 00928-105; 2020-002771-35 (EudraCT Number)
Record Dates: First submitted 2020-10-06; First posted 2020-10-09 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndromes; Multiple Myeloma; Anemia
Keywords: Myelodysplastic Syndromes; Multiple Myeloma; Anemia; LIMBER
MeSH Terms: conditions — Myelodysplastic Syndromes; Multiple Myeloma; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB000928 (Experimental): INCB000928 will be administered in participants with MDS or MM who are transfusion-dependent or present with symptomatic anemia.
  Interventions: Drug: INCB000928

INTERVENTIONS:
Drug: INCB000928 — INCB000928 will be administered once daily.

SUMMARY:
This Phase 1/2, open-label, dose-finding study is intended to evaluate the safety and tolerability, PK, PD, and efficacy of INCB000928 administered as monotherapy in participants with MDS or MM who are transfusion-dependent or present with symptomatic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to avoid pregnancy or fathering children.
* Participants who are transfusion-dependent or present with symptomatic anemia

For MDS participants:

* Ineligible to receive or have not responded to available therapies for anemia such as ESAs or lenalidomide.
* Not requiring cytoreductive therapy other than hydroxyurea.
* BM and peripheral blood myeloblast count < 10%.
* Histologically confirmed diagnosis of the MDS, CMML and unclassifiable MDS/MPN overlap syndromes.

For MM participants:

* Histologically confirmed diagnosis of MM.
* After failure of available standard treatments such as alkylating agents, glucocorticoids, immunomodulatory drugs (lenalidomide,pomalidomide, or thalidomide), proteasome inhibitors (bortezomib or carfilzomib), and daratumumab.

Exclusion Criteria:

* Any prior allogeneic stem cell transplantation or a candidate for such transplantation.
* Any major surgery within 28 days before the first dose of study drug.
* Any prior chemotherapy, immunomodulatory drug therapy, immunosuppressive therapy, biological therapy, endocrine therapy, targeted therapy, or antibody or hypomethylating agent to treat the participant's disease within 5 half-lives or 28 days (whichever is shorter) before the first dose of study drug.
* Undergoing treatment with another investigational medication or having been treated with an investigational medication within 28 days before the first dose of study drug. -Undergoing treatment with ESAs, granulocyte colony-stimulating factor or granulocyte/macrophage colony-stimulating factor, romiplostin, or eltrombopag at any time within 28 days before the first dose of study drug.
* Undergoing treatment with a strong or potent inhibitor or inducer of CYP3A4/5 within 28 days or 5 half-lives (whichever is longer) before the first dose of study drug or expected to receive such treatment during the study.
* History of clinically significant or uncontrolled cardiac disease.
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically Meaningful.
* Presence of chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment.
* Diagnosis of chronic liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekatarine Asatiani, MD, Study Director — Incyte Corporation
Locations (15):
- United States (8):
  - Stanford Cancer Center, Palo Alto, California
  - University of Miami, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Tulane Comprehensive Cancer Center, New Orleans, Louisiana
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
- France (3):
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Italy (4):
  - L Azienda Ospedaliero-Universitaria Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Comitato Di Bioetica Della Fondazione Irccs Policlinico San Matteo, Pavia
  - Irccs Istituto Clinico Humanitas, Rozzano

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 8 study centers in the United States, France, and Italy.
Groups:
- Zilurgisertib 50 mg QD: Participants with myelodysplastic syndromes (MDS) or multiple myeloma (MM) who were transfusion dependent or presented with symptomatic anemia received oral zilurgisertib 50 milligrams (mg) once daily (QD) administered as a monotherapy for up to 6 months.
- Zilurgisertib 100 mg QD: Participants with MDS or MM who were transfusion dependent or presented with symptomatic anemia received oral zilurgisertib 100 mg QD administered as a monotherapy for up to 6 months.
- Zilurgisertib 200 mg QD: Participants with MDS or MM who were transfusion dependent or presented with symptomatic anemia received oral zilurgisertib 200 mg QD administered as a monotherapy for up to 6 months.
- Zilurgisertib 400 mg QD: Participants with MDS or MM who were transfusion dependent or presented with symptomatic anemia received oral zilurgisertib 400 mg QD administered as a monotherapy for up to 6 months.
- Zilurgisertib 600 mg QD: Participants with MDS or MM who were transfusion dependent or presented with symptomatic anemia received oral zilurgisertib 600 mg QD administered as a monotherapy for up to 6 months.
Period: Overall Study
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Started | 4 | 5 | 4 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 4 | 5 | 3
Not completed — Death | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 3 | 2 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1 | 0
Not completed — Participant Started New Therapy; Did Not Return to Clinic | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD | Total
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (4.50) | 74.6 (3.78) | 78.5 (6.19) | 74.8 (4.87) | 75.7 (6.66) | 74.4 (5.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 4 | 1 | 10
  Male | 2 | 4 | 2 | 1 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 5 | 4 | 3 | 3 | 16
  Unknown or Not Reported | 3 | 0 | 0 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 1 | 5 | 3 | 3 | 3 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE is an AE reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 950 days
Population: Full Analysis Set-MDS: all participants with myelodysplastic syndromes (MDS) or MDS/myeloproliferative neoplasm (MPN) overlap syndromes who received at least 1 dose of zilurgisertib
Measure: Count of Participants; unit: Participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 3
Participants | 4 | 5 | 4 | 5 | 2

2. Primary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: The severity of AEs was assessed using Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) Grades 1 through 5. The investigator made an assessment of intensity for each AE and SAE reported during the study and assigned it to one of the following categories. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 950 days
Population: Full Analysis Set-MDS
Measure: Count of Participants; unit: Participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 3
Participants | 2 | 3 | 2 | 2 | 2

3. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any protocol-defined toxicities occurring during the first study drug treatment cycle, from C1D1 up to and including Cycle 1 Day 28 (per regimen cycle schedule), except those with a clear alternative explanation (e.g., disease progression) or transient (≤72 hours) abnormal laboratory values without associated clinically significant signs or symptoms based on investigator determination.
Time Frame: up to Day 28
Population: DLT Evaluable Population: all participants in the FAS Population who met the following criteria: observed for at least the first treatment cycle (i.e., 28 days); received ≥75% of doses of study treatment at the level assigned to that cohort (i.e., 21 days of treatment) or had a DLT during the first study treatment cycle; did not receive any strong or potent CYP3A4/5 inhibitor or inducer during the first study drug treatment cycle (DLT assessment period); was not part of a backfill cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the dose at which the observed DLT rate was closest to the target DLT rate of 28% using an isotonical method that took the assumption of a monotonic dose-toxicity relationship into account. Bayesian optimal interval (BOIN) design was used to determine the MTD for this study. Per the protocol, the stopping rule was either (a) reaching a certain number of participants at one dose level under the early stopping rule or (b) reaching the pre-defined maximum sample size. Dose escalation was to be considered complete only when one of these conditions was met. After completion, the MTD was to be defined as the dose level closest to the target DLT rate. The MTD could not be concluded until the stopping rule was met.
Time Frame: up to Day 28
Population: Full Analysis Set-MDS
Measure: Number; unit: milligrams
Groups:
- All Participants: Participants with MDS or MM who were transfusion dependent or presented with symptomatic anemia received oral zilurgisertib QD administered as a monotherapy for up to 6 months.
Arm/Group | All Participants
Number analyzed (Participants) | 21
milligrams | NA — The maximum sample size for each dose level was 9. Given that there were 2 DLT-evaluable participants at the 600 mg QD dose level and 1 DLT was observed, the dose should have been de-escalated. As a result, the dose escalation was incomplete at the time of study termination, and the MTD could not be determined since the stopping rule had not been met.

5. Primary Outcome: Recommended Dose for Expansion (RDE)
Description: RDE doses were defined as pharmacodynamically active. RDE doses were not to have exceeded the MTD defined in each treatment group.
Time Frame: up to Day 28
Population: Full Analysis Set-MDS
Measure: Number; unit: milligrams
Arm/Group | All Participants
Number analyzed (Participants) | 21
milligrams | NA — The RDE was not established because, at the time of early study termination, dose escalation was ongoing and the dose that had evidence of the best pharmacologic activity while being below the MTD had not yet been identified.

6. Secondary Outcome: Percentage of Participants With Anemia Response
Description: Participants with anemia response were those with a hemoglobin (Hgb) increase of ≥1.5 grams per deciliter (g/dL) relative to baseline for any 8-week period (with each assessment meeting this requirement) during the first 24 weeks of treatment if transfusion independent at baseline. Transfusion-independent participants at baseline were those that did not receive ≥4 units of red blood cell (RBC) transfusions during the 28 days immediately preceding Cycle 1 Day 1 or did not receive ≥4 units of RBC transfusions in the 8 weeks immediately preceding Cycle 1 Day 1, for an Hgb level of <8.5 g/dL, in the absence of bleeding or treatment-induced anemia.
Time Frame: up to Week 24
Population: Full Analysis Set-MDS. Participants must have been on treatment for ≥8 consecutive weeks or discontinued treatment before Week 8. Only participants who were transfusion independent at baseline were analyzed. The 95% confidence interval was calculated using exact binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 2 | 4 | 2 | 4 | 2
percentage of participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 84.2]

7. Secondary Outcome: Duration of Anemia Response
Description: Duration of anemia response was defined as the interval from the first onset of anemia response to the earliest date of loss of anemia response that persisted for at least 4 weeks or death from any cause. Participants with anemia response were those with a hemoglobin (Hgb) increase of ≥1.5 grams per deciliter (g/dL) relative to baseline for any 8-week period (with each assessment meeting this requirement) during the first 24 weeks of treatment if transfusion independent at baseline. Transfusion-independent participants at baseline were those that did not receive ≥4 units of red blood cell (RBC) transfusions during the 28 days immediately preceding Cycle 1 Day 1 or did not receive ≥4 units of RBC transfusions in the 8 weeks immediately preceding Cycle 1 Day 1, for an Hgb level of <8.5 g/dL, in the absence of bleeding or treatment-induced anemia.
Time Frame: up to 920 days
Population: Full Analysis Set-MDS. Participants must have been on treatment for ≥8 consecutive weeks and have discontinued treatment before Week 8. Only participants who were transfusion independent at baseline and had a response were analyzed.
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With RBC-transfusion Independence (TI)
Description: Participants with RBC-transfusion independence were defined as those who did not require any RBC transfusion for at least 8 consecutive weeks during the first 24 weeks of treatment.
Time Frame: up to Week 24
Population: Full Analysis Set-MDS. Only participants who were transfusion dependent at Baseline were analyzed. The 95% confidence interval was calculated using exact binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1
percentage of participants | 0.0 [0.0 to 84.2] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]

9. Secondary Outcome: Duration of RBC-transfusion Independence (TI) Period for Participants Achieving RBC-TI for at Least 8 Consecutive Weeks During the First 24 Weeks of Treatment
Description: Participants with RBC-TI were defined as those who did not require any RBC transfusion for at least 8 consecutive weeks during the first 24 weeks of treatment.
Time Frame: up to 920 days
Population: Full Analysis Set-MDS. Only participants who were transfusion dependent at Baseline and achieved transfusion independence were analyzed.
Measure: Median (Standard Error); unit: days
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
days |  | 60 (NA) — Standard error cannot be calculated for a single participant. |  |  |

10. Secondary Outcome: Rate of Red Blood Cell (RBC) Transfusion From Week 12 Through Week 24
Description: The rate of RBC transfusion was defined as the average number of RBC units per participant-month during the treatment period.
Time Frame: from Week 12 through Week 24
Population: Full Analysis Set-MDS. Only participants who were on treatment for at least 78 days were included in the analysis.
Measure: Mean (Standard Deviation); unit: RBC units per participant-month
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 3
RBC units per participant-month | 2.53 (1.955) | 1.34 (0.948) | 3.01 (2.955) | 2.71 (2.232) | 1.19 (2.067)

11. Secondary Outcome: The Largest Increase From Baseline in the Mean Hgb Values Over Any Rolling 8-week Treatment Period During the First 24 Weeks of Treatment
Description: Baseline Hgb was measured up to 8 weeks prior to the first dose administration of zilurgisertib. The baseline Hgb was defined as the average of all eligible Hgb assessments. The Hgb assessment(s) within the window from the date received RBC transfusion+1 day to the date received RBC transfusion+14 days that didn't trigger another transfusion were excluded.
Time Frame: up to Week 24
Population: Full Analysis Set-MDS. Participants were included in the mean change from baseline in hemoglobin value analysis if the participant was in the FAS and met both of the following criteria: a. was on treatment for more than 8 weeks; b. had ≥1 valid post-baseline Hgb assessment(s).
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
grams per liter | 2.19 (2.782) | 9.73 (2.842) | 2.51 (3.681) | 4.92 (10.240) | 6.59 (4.229)

12. Secondary Outcome: Overall Response Rate (ORR) in MDS Participants
Description: ORR was defined as the percentage of participants with complete response (CR) or partial response (PR). For MDS, CR: bone marrow with ≤5% myeloblasts with normal maturation of all cell lines; HgB ≥11 g/dl, neutrophils ≥1.0x10^9/Liter (L), platelets ≥100x10^9/L, and no blasts in the peripheral blood. For MDS, PR: all CR criteria, but bone marrow blasts decreased by ≥50% over pretreatment but still >5%; cellularity and morphology not relevant. For MDS/MPN overlap syndromes, CR: bone marrow with ≤5% myeloblasts; no osteomyelofibrosis or ≤Grade 1 fibrosis; white blood cells ≤10X10^9 cells/L, HgB ≥11 g/dL, platelets ≥100x10^9/L/≤450x10^9/L, neutrophils ≥1.0x10^9/L, no blasts, neutrophil precursors reduced to ≤2%, monocytes ≤1x10^9/L in peripheral blood; complete resolution of medullary disease. For MDS/MPN overlap syndromes, PR: normalization of peripheral counts and hepatosplenomegaly with bone marrow blasts reduced by 50%, but remaining >5% of cellularity.
Time Frame: up to 920 days
Population: Full Analysis Set-MDS only. Participants with MDS/MPN overlap syndromes were excluded from analysis. The 95% confidence interval was calculated using exact binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 3
percentage of participants | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8]

13. Secondary Outcome: Percentage of MDS Participants With an Event of Progression or Death
Description: Participants with MDS/MPN overlap syndromes were excluded from analysis. Data have been reported as the percentage of participants with an event of progression or death rather than median PFS (the interval from the first dose of study drug until the first documented progression or death) because 2 participants had an event of PFS or death. It was pre-specified in the SAP that the number of MDS participants with documented progression or death was to be summarized.
Time Frame: up to 920 days
Population: Full Analysis Set-MDS only. Participants with MDS/MPN overlap syndromes were excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 3
percentage of participants | 25.0 | 0.0 | 0.0 | 20.0 | 0.0

14. Secondary Outcome: Percentage of Participants With an Event of Leukemia or Death
Description: Data have been reported as the percentage of participants with an event of leukemia or death rather than LFS (the interval from the first dose of study drug until the first documented leukemia transformation or death from any cause) because 3 participants had an event of leukemia or death. It was pre-specified in the SAP that the number of participants with leukemia transformation or death was to be summarized.
Time Frame: up to 920 days
Population: Full Analysis Set-MDS
Measure: Number; unit: percentage of participants
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 3
percentage of participants | 25.0 | 20.0 | 0.0 | 20.0 | 0.0

15. Secondary Outcome: ORR in Multiple Myeloma (MM) Participants
Description: ORR was defined as the percentage of participants with stringent CR, CR, very good PR, and PR.
Time Frame: up to 920 days
Population: Full Analysis Set. No participants with MM were enrolled.
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: PFS in MM Participants
Description: PFS was defined as the interval from the first dose of study drug until the first documented progression or death.
Time Frame: up to 920 days
Population: Full Analysis Set. No participants with MM were enrolled.
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Cmax of Zilurgisertib
Description: Cmax was defined as the maximum concentration of zilurgisertib.
Time Frame: Days 1 and 15 of Cycle 1: pre-dose; 2, 4, and 6 hours post-dose
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of zilurgisertib and provided at least 1 postdose plasma sample (1 PK measurement). Only participants with available data were analyzed. One participant who was supposed to receive 100 mg actually received 25 mg from Day 1 to Day 16.
Measure: Mean (Standard Deviation); unit: nanomolar
Groups:
- Zilurgisertib 25 mg QD: Participants with myelodysplastic syndromes (MDS) or multiple myeloma (MM) who were transfusion dependent or presented with symptomatic anemia received oral zilurgisertib 25 milligrams (mg) once daily (QD) administered as a monotherapy from Day 1 to Day 16.
Arm/Group | Zilurgisertib 25 mg QD | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 1 | 4 | 4 | 4 | 4 | 2
nanomolar
  Cycle 1 Day 1 | 79.9 (NA) — Standard deviation was not calculated for a single participant. | 181 (80.4) | 249 (100) | 569 (291) | 1950 (652) | NA (NA) — Two participants had values above the upper limit of quantification, meaning data for PK parameters could not be determined.
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2 | 2
  Cycle 1 Day 15 |  | 350 (131) | 636 (330) | 1360 (613) | 2620 (4620) | NA (NA) — Two participants had values above the upper limit of quantification, meaning data for PK parameters could not be determined.

18. Secondary Outcome: Tmax of Zilurgisertib
Description: tmax was defined as the time to the maximum observed concentration of zilurgisertib.
Time Frame: Days 1 and 15 of Cycle 1: pre-dose; 2, 4, and 6-8 hours post-dose
Population: PK Evaluable Population. Only participants with available data were analyzed. One participant who was supposed to receive 100 mg actually received 25 mg from Day 1 to Day 16.
Measure: Median (Full Range); unit: hours
Arm/Group | Zilurgisertib 25 mg QD | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 1 | 4 | 4 | 4 | 4 | 2
hours
  Cycle 1 Day 1 | 2.0 [NA to NA] — Min, max are not reported for a single participant. | 2.0 [2.0 to 4.0] | 2.0 [2.0 to 2.0] | 3.0 [2.0 to 4.0] | 2.0 [2.0 to 2.0] | NA [NA to NA] — Two participants had values above the upper limit of quantification, meaning data for PK parameters could not be determined.
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2 | 2
  Cycle 1 Day 15 |  | 2.0 [2.0 to 6.0] | 2.0 [2.0 to 2.0] | 3.0 [2.0 to 6.0] | 2.0 [2.0 to 4.0] | NA [NA to NA] — Two participants had values above the upper limit of quantification, meaning data for PK parameters could not be determined.

19. Secondary Outcome: AUClast of Zilurgisertib
Description: AUClast was defined as the area under the plasma concentration-time curve from time 0 to the last quantifiable measurable plasma concentration of zilurgisertib.
Time Frame: Days 1 and 15 of Cycle 1: pre-dose; 2, 4, and 6-8 hours post-dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanomolar x hour
Arm/Group | Zilurgisertib 25 mg QD | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 1 | 4 | 4 | 4 | 4 | 2
nanomolar x hour
  Cycle 1 Day 1 | 343 (NA) — Standard deviation was not calculated for a single participant. | 749 (312) | 1070 (471) | 2540 (1150) | 8050 (2680) | NA (NA) — Two participants had values above the upper limit of quantification, meaning data for PK parameters could not be determined.
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2 | 2
  Cycle 1 Day 15 |  | 1890 (749) | 3090 (1620) | 6850 (3050) | 12300 (26100) | NA (NA) — Two participants had values above the upper limit of quantification, meaning data for PK parameters could not be determined.

20. Secondary Outcome: Ctrough of Zilurgisertib
Description: Ctrough was defined as the lowest concentration of zilurgisertib.
Time Frame: Day 15 of Cycle 1: pre-dose; 2, 4, and 6-8 hours post-dose
Population: PK Evaluable Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanomolar
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 2
nanomolar | 214 (91.8) | 304 (175) | 619 (241) | 981 (3130) | NA (NA) — Two participants had values above the upper limit of quantification, meaning data for PK parameters could not be determined.

21. Secondary Outcome: Percentage Change in Hepcidin From Cycle 1 Day 15 to Cycle 7 Day 1
Description: Percentage change was calculated as the ([post-baseline value minus the baseline value] / [baseline value]) * 100.
Time Frame: from Cycle 1 Day 15 to Cycle 7 Day 1
Population: Pharmacodynamic (PD) Evaluable Population: all participants who received at least 1 dose of zilurgisertib and provided at least 1 plasma/serum sample (1 PD measurement)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 3
percent change | -24.53 (41.69) | -16.25 (47.06) | -11.25 (39.97) | -59.02 (32.35) | -63.79 (44.23)

22. Secondary Outcome: Change From Baseline in Ferritin
Description: Change from Baseline (CFB) was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Cycle 1 Day 8; Cycle 1 Day 15; Cycles 2, 3, 4, 5, 6, and 7 Day 1
Population: Full Analysis Set-MDS. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 3
nanograms per milliliter
  Baseline | 1022.35 (634.096) | 930.18 (697.078) | 2092.25 (1220.166) | 2034.42 (1329.794) | 1469.00 (1191.873)
  CFB at Cycle 1 Day 8: number analyzed (Participants) | 3 | 5 | 4 | 3 | 2
  CFB at Cycle 1 Day 8 | 47.67 (43.501) | -65.24 (57.388) | 203.25 (523.789) | -98.83 (567.584) | -110.00 (24.042)
  CFB at Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 4 | 3 | 2
  CFB at Cycle 1 Day 15 | 292.00 (161.220) | 17.30 (31.109) | 67.50 (140.950) | -109.77 (98.223) | -96.00 (56.569)
  CFB at Cycle 2 Day 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 2
  CFB at Cycle 2 Day 1 | 101.65 (245.814) | 70.03 (76.619) | 154.50 (453.658) | -92.87 (364.312) | 135.00 (200.818)
  CFB at Cycle 3 Day 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
  CFB at Cycle 3 Day 1 | 307.58 (709.602) | -6.70 (46.054) | 532.00 (833.804) | 353.77 (314.682) | -383.00 (536.324)
  CFB at Cycle 4 Day 1: number analyzed (Participants) | 3 | 2 | 4 | 5 | 2
  CFB at Cycle 4 Day 1 | 409.83 (689.052) | -21.15 (48.295) | 875.00 (649.850) | 619.00 (275.281) | -153.50 (82.731)
  CFB at Cycle 5 Day 1: number analyzed (Participants) | 3 | 1 | 4 | 4 | 2
  CFB at Cycle 5 Day 1 | 349.00 (680.559) | 172.00 (NA) — Standard deviation was not calculated for a single participant. | 574.00 (394.335) | 516.10 (502.323) | -106.50 (211.425)
  CFB at Cycle 6 Day 1: number analyzed (Participants) | 3 | 2 | 3 | 2 | 0
  CFB at Cycle 6 Day 1 | 297.67 (614.180) | 488.50 (152.028) | 347.33 (362.417) | 442.15 (264.246) |
  CFB at Cycle 7 Day 1: number analyzed (Participants) | 2 | 1 | 3 | 2 | 0
  CFB at Cycle 7 Day 1 | 365.50 (658.316) | 971.00 (NA) — Standard deviation was not calculated for a single participant. | 315.33 (222.172) | 507.35 (64.559) |

23. Secondary Outcome: Change From Baseline in Hemoglobin at the End of Treatment
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: up to 950 days
Population: Full Analysis Set-MDS. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 3
grams per liter
  Baseline | 77.7750 (5.83688) | 75.7200 (4.00899) | 74.9354 (5.98330) | 74.6767 (7.94708) | 79.4139 (4.14997)
  Change from Baseline at end of treatment: number analyzed (Participants) | 2 | 3 | 2 | 3 | 3
  Change from Baseline at end of treatment | -1.7500 (4.59619) | 10.1333 (12.87685) | 4.0182 (7.61104) | 16.9556 (12.34055) | 69.6667 (10.40833)

ADVERSE EVENTS:
Time Frame: up to 950 days
Description: Analysis was conducted in the Full Analysis Set-MDS, comprised of all participants with myelodysplastic syndromes (MDS) or MDS/myeloproliferative neoplasm (MPN) overlap syndromes who received at least 1 dose of zilurgisertib.
Groups:
- Total: Total
Arm/Group | Zilurgisertib 50 mg QD | Zilurgisertib 100 mg QD | Zilurgisertib 200 mg QD | Zilurgisertib 400 mg QD | Zilurgisertib 600 mg QD | Total
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/5 | 0/4 | 1/5 | 0/3 | 3/21
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/5 | 2/4 | 2/5 | 0/3 | 7/21
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 4/4 | 5/5 | 2/3 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilurgisertib 50 mg QD (N=4) | Zilurgisertib 100 mg QD (N=5) | Zilurgisertib 200 mg QD (N=4) | Zilurgisertib 400 mg QD (N=5) | Zilurgisertib 600 mg QD (N=3) | Total (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilurgisertib 50 mg QD (N=4) | Zilurgisertib 100 mg QD (N=5) | Zilurgisertib 200 mg QD (N=4) | Zilurgisertib 400 mg QD (N=5) | Zilurgisertib 600 mg QD (N=3) | Total (N=21)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Amylase increased (Investigations) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 3 (5)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bankart lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Malaise (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 6 (6)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 4 (6)
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The sponsor terminated study enrollment as a strategic decision. Due to early study termination, no participants were enrolled in the expansion stage of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT04582539/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT04582539/SAP_001.pdf